CLINICAL TRIAL: NCT07304999
Title: Surgical and Audiological Outcomes of Endoscopic Stapes Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Sayed Abdelrahman, Specialist department TemaGeneral hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-11-2MD
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Otosclerosis
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endsocopic stapedotomy — Patients will undergo stapedotomy by endoscopic approach and the same type of artificial loop prosthesis will be used .
  Intraoperative details are recorded including invasiveness of the surgery, clarity of the exposure of the middle ear and stapedial structures , the ease of placement of the artificial loop prosthesis and also intraoperative complications.
  Postoperative follow up and complications will be recorded and evaluated. Postoperative audiological evaluation, including air-conduction (AC), bone-conduction (BC) and air-bone gap (ABG), will be carried out using pure-tone audiometry and performed within 4 to 6 months after surgery.

SUMMARY:
Otosclerosis is a pathological bone remodeling process that affects the middle and inner ears. It was first reported by Antonio Maria Valsalva in 1735 and subsequently described pathologically by Adam Politzer in 1839 .

In otosclerosis, the normal, dense endochondral bone of the otic capsule around the inner ear labyrinth is replaced by irregularly laid spongy bone, which subsequently hardens and leads to fixation of the stapes footplate . Otosclerosis causes progressive conductive hearing loss that typically presents with a normal tympanic membrane. However, a reddish shadow on the promontory of the cochlea may be seen in some cases (Schwartze sign) if the tympanic membrane is clear enough.

Initial symptoms of otosclerosis include decreased sensitivity to low-frequency sounds, such as whispers. Patients may also paradoxically deny difficulty hearing conversation in loud background noise, which is termed "paracusis Willisii" or "paracusis of Willis,. Tinnitus may worsen as the disease progresses. Vertigo is usually mild, but as the disease progresses, balance may deteriorate, mimicking Ménière disease. .

On physical examination, patients with otosclerosis may speak in low volume and monotonous voices. Otoscopy may reveal no abnormalities at all. With active otosclerosis, however, increased vascularity of the cochlear promontory may be visible through the tympanic membrane A Weber test performed with a 512 Hz (Hertz) fork will generally lateralize toward the ear with the conductive loss or toward the ear with the greater conductive loss in cases of bilateral otosclerosis . In most cases of otosclerosis, pure tone audiometry shows low frequency decreases in air conduction thresholds. Bone conduction, however, typically remains normal. A "Carhart notch" is often seen, which is an artifactual dip in the bone conduction line by 20-30 dB(disciple) at 2,000 Hz due to the resonance frequency of the ossicular chain .

There is no medical therapy that is curative for otosclerosis. Though sodium fluoride is prescribed to slow the progression of otosclerosis, its efficacy is still controversial and In stapes surgery different surgical techniques, approaches and prostheses in order to restore sound transmission have been described. Stapedectomy was first described by Shea.Jr in 1956.

Surgical techniques for treatment of otosclerosis have been improved, updated, or adjusted over time to lower intraoperative and post-operative problems and boost overall effectiveness .

The treatment of choice is stapedotomy or stapedectomy, along with the placement of a prosthesis. In these procedures, either a hole is drilled in the center of the stapes footplate with a high-speed microdrill or a laser (stapedotomy), and a prosthesis is placed between the long process of the incus and the oval window membrane via the hole in the stapes footplate, or the stapes footplate is removed partially or in its entirety and a prosthesis placed between the incus and the oval window, typically with a vein or fascia graft used to protect the oval window membrane (stapedectomy). In both procedures, the crura of the stapes are fractured, and the incudo stapedial joint is divided in order to permit the removal of the stapes superstructure.

Surgical treatment for otosclerosis generally produces good outcomes, irrespective of the approach employed, provided appropriate patient selection. For patients with bilateral otosclerosis, the ear with greater hearing loss is typically addressed first; both ears are not operated under the same anesthetic in order to avoid the very unlikely scenario in which total sensorineural hearing loss occurs bilaterally as a result of surgery. A 2018 review published by Cheng et al indicated comparable results between stapedotomy and stapedectomy, with a slight advantage in terms of high- frequency hearing and complication rate for stapedotomy .

Microscopic trans canal or end aural approach is the most preferred technique in stapes surgery . Although microscopes provide good magnification and let both hands use, sufficient exposure of stapedial structures might not be possible under microscopic approach without bone curettage .

In microscopic approaches, extensive curettage of scutum may result in complications such as chorda tympani nerve injury, impaired taste sensation, subluxation of ossicles, retraction pockets and postoperative higher pain levels .

ELIGIBILITY:
Inclusion Criteria:

* Patients with otosclerosis who will undergo endoscopic stapedotomy whose diagnoses are mainly based on progressive conductive deafness over 25 dB in the range of 0.25-4 kHz.

Exclusion Criteria:

* Otosclerotic patients with either isolated sensorineural or mixed deafness (bone conduction more than 30 dB), or those with small air-bone gap less than 25 dB and those complaining from vestibular symptoms in the last year prior to surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
hearing level | 6 monthes
  changes in air-bone gap(by decibles) by using pure tone audiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag universty hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quinn KJ, Coelho DH. The Curious Rise and Incomplete Fall of "Paracusis Willisii". Otol Neurotol. 2022 Jan 1;43(1):137-143. doi: 10.1097/MAO.0000000000003368. PMID 34619730
- [Background] Kelly EA, Li B, Adams ME. Diagnostic Accuracy of Tuning Fork Tests for Hearing Loss: A Systematic Review. Otolaryngol Head Neck Surg. 2018 Aug;159(2):220-230. doi: 10.1177/0194599818770405. Epub 2018 Apr 17. PMID 29661046
- [Background] Cheng HCS, Agrawal SK, Parnes LS. Stapedectomy Versus Stapedotomy. Otolaryngol Clin North Am. 2018 Apr;51(2):375-392. doi: 10.1016/j.otc.2017.11.008. Epub 2018 Feb 3. PMID 29397948
- [Background] Hoskison EE, Harrop E, Jufas N, Kong JHK, Patel NP, Saxby AJ. Endoscopic Stapedotomy: A Systematic Review. Otol Neurotol. 2021 Dec 1;42(10):e1638-e1643. doi: 10.1097/MAO.0000000000003242. PMID 34267093